CLINICAL TRIAL: NCT05956353
Title: Stories for Change: Early Detection Can Save Lives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark L Wieland, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 23-001860
Record Dates: First submitted 2023-06-27; First posted 2023-07-21 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stories for Change: Prevention (S4C) intervention (Experimental): Participants who are due or overdue for cancer screening will receive the digital storytelling intervention and complete a cross-sectional survey to assess intervention acceptability, socio-behavioral constructs, and theory-based constructs.
  Interventions: Behavioral: Digital Storytelling Intervention

INTERVENTIONS:
Behavioral: Digital Storytelling Intervention — Culturally tailored narrative-based videos created by individuals to promote colorectal, breast and cervical cancer screening among eligible participants in a primary care practice.

SUMMARY:
The purpose of this study is to evaluate the Stories for Change (S4C) Cancer Prevention digital storytelling intervention for acceptability and socio-behavioral constructs to increase cancer screening among Hispanic or Latino individuals.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic, Latino/a/x/e, or Chicano/a/x;
* For breast cancer screening: age 40-74 years; for cervical cancer screening: age 21-65 years; for colorectal cancer screening: age 45-75 year
* Receive primary care at either Hennepin Healthcare (HH) or Mountain Park Health Center (MPHC), or Mayo Clinic.
* At least one office visit within the previous 12 months to the primary care site.
* Eligibility for breast, cervical, or colorectal cancer screening documented in the electronic medical record (EMR).
* Intention to continue to receive medical care at HH, MPHC or Mayo Clinic for the next three months.

If a potential participant is eligible for more than one screening, they will be given the option of participating in multiple versions of the intervention.

Exclusion Criteria:

* Individuals with previous breast, cervical, or colorectal cancer diagnoses.
* For the participants in the colorectal cancer screening intervention, those under surveillance (i.e., did not have a cancer diagnosis but did have polyps) will also be excluded.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Number of participants screened and recruited | 1 year
  Our primary measure is the number of participants screened and recruited. We need this information to calculate the number needed to screen in order to recruit one participant from each site in our future randomized controlled trial.

SECONDARY OUTCOMES:
Constructs associated with effective implementation research | 1 year
  Our secondary measure will utilize the Consolidated Framework for Implementation Research. We need this information to identify recruitment successes and opportunities for change in our future randomized controlled trial.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Weiland, MD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Moutain Park Health Center, Phoenix, Arizona
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Mayo Clinic Minnesota, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials